CLINICAL TRIAL: NCT00948324
Title: Effect of Intensive Therapy Associated With CSII on β-cell Function With Newly Diagnosed Type 2 Diabetes
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanbing Li, Department of Endocrinology and Diabetes Center, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, P. R. China, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87755766
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: ype 2 diabetes mellitus, continuous subcutaneous insulin infusion,; α-lipoic acid ,rosiglitazone ,metformin，therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CSII (Active Comparator): CSII: Patients in continuous subcutaneous insulin infusion group received insulin analogue with an insulin pump along.
  Interventions: Drug: CSII,ALA,MET,RSG
- ALA (Active Comparator): ALA:CSII combined with two weeks α- thioctic acid (600mg/500ml NaCl, 0.9%), ivdrip QD.
  Interventions: Drug: CSII,ALA,MET,RSG
- RSG (Active Comparator): RSG:CSII combined with three months rosiglitazoneor 4mg QD.
  Interventions: Drug: CSII,ALA,MET,RSG
- MET (Active Comparator): MET:CSII combined with metformin 500mg BID-TID.
  Interventions: Drug: CSII,ALA,MET,RSG

INTERVENTIONS:
Drug: CSII,ALA,MET,RSG — CSII along.ALA:CSII combined with two weeks α- thioctic acid (600mg/500ml NaCl, 0.9%), ivdrip QD. RSG:CSII combined with three months rosiglitazoneor 4mg QD. MET:CSII combined with metformin 500mg BID-TID.

SUMMARY:
The purpose of this study is to investigate and evaluate the effects of different interventions (1.continuous subcutaneous insulin infusion,2.continuous subcutaneous insulin infusion combined with rosiglitazone 3.continuous subcutaneous insulin infusion combined with metformin,4.continuous subcutaneous insulin infusion combined with α- thioctic acid daily injections,) on glycemic control, B-cell function and the remission rate in newly-diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes,

Exclusion Criteria:

* received previous antihyperglycaemic therapy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2019-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
beta cell function;fast blood glucose; | 2011/05

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan Bing, MD, Principal Investigator — Ministry of Education

REFERENCES:
- [Derived] Liu L, Ke W, Wan X, Zhang P, Cao X, Deng W, Li Y. Insulin requirement profiles of short-term intensive insulin therapy in patients with newly diagnosed type 2 diabetes and its association with long-term glycemic remission. Diabetes Res Clin Pract. 2015 May;108(2):250-7. doi: 10.1016/j.diabres.2015.02.011. Epub 2015 Feb 21. PMID 25765670